CLINICAL TRIAL: NCT01518062
Title: Dose Response Trial of Biosynthetic Authentic Human Growth Hormone and Induction of Puberty With 17b Oestradiol in Girls With Turner's Syndrome
Brief Title: Safety of Somatropin and Induction of Puberty With 17-beta-oestradiol in Girls With Turner Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHTUR/BPD/5-13
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Genetic Disorder; Turner Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome | interventions — Human Growth Hormone; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (Experimental)
  Interventions: Drug: somatropin; Drug: oestrogen
- Medium dose (Experimental)
  Interventions: Drug: somatropin; Drug: oestrogen
- High dose (Experimental)
  Interventions: Drug: somatropin; Drug: oestrogen

INTERVENTIONS:
Drug: somatropin — 4 IU/m^2 body surface for 4 years (main period). In extension period subjects continue the reached dose until final height. Administered as once daily subcutaneous injection
  Arms: Low dose
Drug: somatropin — Initial dose 4 IU/m^2 body surface the first year, then 6 IU/m^2 body surface for 3 years (main period). In extension period subjects continue the reached dose until final height. Administered as once daily subcutaneous injection
  Arms: Medium dose
Drug: somatropin — Initial dose 4 IU/m^2 body surface the first year, then 6 IU/m^2 body surface, the second year and finally 8 IU/m^2 body surface for 2 years (main period). In extension period subjects continue the reached dose until final height. Administered as once daily subcutaneous injection
  Arms: High dose
Drug: oestrogen — Treatment with oestrogen was administered if spontaneous puberty had not occurred by age 12 years and was initiated in the extension period after at least four years of somatropin treatment

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to assess whether increasing doses of somatropin (Norditropin®) can maintain the initial increase in height velocity and improve final height. This trial has two trial periods, a main period of 4 years and an extension period until final height is reached.

ELIGIBILITY:
Inclusion Criteria:

* Turner Syndrome
* Well documented growth rate during the previous year
* Height below the 50th percentile for the age in Dutch children
* Normal thyroid function

Exclusion Criteria:

* Any endocrine or metabolic disorder
* Growth failure due to disorders of genitourinary, cardio-pulmonary, gastro-intestinal and nervous systems, nutritional/vitamins deficiencies and chondrodysplasias
* Patients with hydrocephalus

Ages: 2 Years to 11 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 1989-11; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Final height

SECONDARY OUTCOMES:
Height velocity (cm/year)
Ratio between change in bone age and change in chronological age
Age at onset of puberty
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands

REFERENCES:
- [Result] van Teunenbroek A, de Muinck Keizer-Schrama SM, Stijnen T, Jansen M, Otten BJ, Delemarre-van de Waal HA, Vulsma T, Wit JM, Rouwe CW, Reeser HM, Gosen JJ, Rongen-Westerlaken C, Drop SL. Yearly stepwise increments of the growth hormone dose results in a better growth response after four years in girls with Turner syndrome. Dutch Working Group on Growth Hormone. J Clin Endocrinol Metab. 1996 Nov;81(11):4013-21. doi: 10.1210/jcem.81.11.8923853.
- [Result] Sas TC, Gerver WJ, de Bruin R, Stijnen T, de Muinck Keizer-Schrama SM, Cole TJ, van Teunenbroek A, Drop SL. Body proportions during long-term growth hormone treatment in girls with Turner syndrome participating in a randomized dose-response trial. J Clin Endocrinol Metab. 1999 Dec;84(12):4622-8. doi: 10.1210/jcem.84.12.6225. PMID 10599729
- [Result] Sas TC, Cromme-Dijkhuis AH, de Muinck Keizer-Schrama SM, Stijnen T, van Teunenbroek A, Drop SL. The effects of long-term growth hormone treatment on cardiac left ventricular dimensions and blood pressure in girls with Turner's syndrome. Dutch Working Group on Growth Hormone. J Pediatr. 1999 Oct;135(4):470-6. doi: 10.1016/s0022-3476(99)70170-8. PMID 10518081
- [Result] Van Pareren YK, De Muinck Keizer-Schrama SM, Stijnen T, Sas TC, Drop SL. Effect of discontinuation of long-term growth hormone treatment on carbohydrate metabolism and risk factors for cardiovascular disease in girls with Turner syndrome. J Clin Endocrinol Metab. 2002 Dec;87(12):5442-8. doi: 10.1210/jc.2002-020789. PMID 12466334
- [Result] van Pareren YK, de Muinck Keizer-Schrama SM, Stijnen T, Sas TC, Jansen M, Otten BJ, Hoorweg-Nijman JJ, Vulsma T, Stokvis-Brantsma WH, Rouwe CW, Reeser HM, Gerver WJ, Gosen JJ, Rongen-Westerlaken C, Drop SL. Final height in girls with turner syndrome after long-term growth hormone treatment in three dosages and low dose estrogens. J Clin Endocrinol Metab. 2003 Mar;88(3):1119-25. doi: 10.1210/jc.2002-021171. PMID 12629094
- [Result] van Pareren YK, Duivenvoorden HJ, Slijper FM, Koot HM, Drop SL, de Muinck Keizer-Schrama SM. Psychosocial functioning after discontinuation of long-term growth hormone treatment in girls with Turner syndrome. Horm Res. 2005;63(5):238-44. doi: 10.1159/000085841. Epub 2005 May 17. PMID 15900109
- [Result] Sas TC, de Muinck Keizer-Schrama SM, Stijnen T, Jansen M, Otten BJ, Hoorweg-Nijman JJ, Vulsma T, Massa GG, Rouwe CW, Reeser HM, Gerver WJ, Gosen JJ, Rongen-Westerlaken C, Drop SL. Normalization of height in girls with Turner syndrome after long-term growth hormone treatment: results of a randomized dose-response trial. J Clin Endocrinol Metab. 1999 Dec;84(12):4607-12. doi: 10.1210/jcem.84.12.6241. PMID 10599727
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com